CLINICAL TRIAL: NCT04793139
Title: Efficacy and Safety of Camrelizumab for Chinese NSCLC Patients: a Prospective, Observational, Multicenter Real-World Study
Brief Title: Efficacy and Safety of Camrelizumab in Real-World Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CTONG2007
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab-treated advanced NSCLC Patients with advanced non-small cell lung cancer treated with camrelizumab. Dosage form, dosage, frequency and duration of camrelizumab is determined according to the investigator's actual clinical practice.
  Other Names: SHR-1210

SUMMARY:
This observational real-world study is designed to evaluate the efficacy and safety of camrelizumab for the treatment of Chinese NSCLC patients.

DETAILED DESCRIPTION:
Camrelizumab is a humanized antibody for cancer immunotherapy. The National Medical Products Administration (NMPA, China) approved camrelizumab as a first-line treatment of certain patients with NSCLC. This is a multicenter non-interventional study, NSCLC patients who have been treated with camrelizumab will be included. The main objective of this study is to evaluate the efficacy and safety of camrelizumab in the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent and volunteer to participate in the study;
2. Non-small cell lung cancer confirmed by histological/cytopathological tests;
3. Age ≥18;
4. The investigators determined that patients should receive camrelizumab alone or in combination.

Exclusion Criteria:

1. Patients who are also receiving other immunomedications or therapies;
2. Patients participating in other interventional studies;
3. Patients complicated with other malignant tumors;
4. Women who have been confirmed to be pregnant or lactating;
5. The Investigator considers the patient unsuitable for participation in any other condition of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total 1000 patients who should accept camrelizumab with NSCLC will be enrolled. The patients should be registered consecutively in each site.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
AE,Grade 3-5 | From April 1, 2021 to Septeember 30, 2024
  Safety of the general population:Serious Adverse Events (AE)，Grade 3-5.

SECONDARY OUTCOMES:
pCR | From April 1, 2021 to December 30, 2024
  Neoadjuvant therapy population: pathological complete response rate (pCR).
MPR | From April 1, 2021 to December 30, 2024
  Neoadjuvant population: main pathological response rate (MPR)
R0 resection rate | From April 1, 2021 to December 30, 2022
  Neoadjuvant therapy population: R0 resection rate.
ORR | From April 1, 2021 to December 30, 2022
  Advanced non-small cell lung cancer: objective response rate (ORR).
PFS | From April 1, 2021 to December 30, 2022
  Advanced non-small cell lung cancer: progression-free survival.
OS | From April 1, 2021 to December 30, 2022
  Advanced non-small cell lung cancer: Overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, Principal Investigator — Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided